CLINICAL TRIAL: NCT01508910
Title: A Prospective, Randomized, Double-blinded, Active-control and Unblinded Standard of Care (SOC) Controlled Study to Determine the Efficacy and Safety of Targeted Intramyocardial Delivery of Autologous CD34+ Cells (Auto-CD34+ Cells) for Increasing Exercise Capacity During Standardized Exercise Testing in Subjects With Refractory Angina Pectoris and Chronic Myocardial Ischemia
Brief Title: Efficacy and Safety of Targeted Intramyocardial Delivery of Auto CD34+ Stem Cells for Improving Exercise Capacity in Subjects With Refractory Angina
Acronym: RENEW
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lisata Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 901001; RENEW Study (Other: Caladrius Biosciences, Inc.)
Record Dates: First submitted 2012-01-10; First posted 2012-01-12 (Estimated); Results first posted 2017-02-15 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Chronic Myocardial Ischemia; Refractory Angina Pectoris; Advanced Coronary Heart Disease
MeSH Terms: conditions — Angina Pectoris | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Treatment Arm (Experimental): Targeted intramyocardial delivery of 1 x 10^5 Auto-CD34+ cells after granulocyte-colony stimulating factor (G-CSF) mobilization and apheresis
  Interventions: Biological: Auto-CD34+ cells
- Active Control Arm (Placebo Comparator): Targeted intramyocardial delivery of placebo after G-CSF mobilization and apheresis
  Interventions: Biological: Placebo: Diluent used to suspend Auto-CD34+ cells
- Unblinded Standard of Care (SOC) Arm (Other): No study-related procedures will be performed.
  Interventions: Other: Standard of care

INTERVENTIONS:
Biological: Auto-CD34+ cells — 10 intramyocardial injections of 0.2 mL per injection site of Auto-CD34+ cells
  Arms: Treatment Arm
Biological: Placebo: Diluent used to suspend Auto-CD34+ cells — 10 intramyocardial injections of 0.2 mL per injection site of placebo
  Arms: Active Control Arm
Other: Standard of care — Standard of care for refractory angina
  Arms: Unblinded Standard of Care (SOC) Arm

SUMMARY:
The purpose of the study is to assess the safety and efficacy of targeted intramyocardial delivery of Auto-CD34+ cells for increasing exercise time and amelioration of anginal symptoms in subjects with refractory angina and chronic myocardial ischemia.

ELIGIBILITY:
Main Inclusion Criteria:

* Male or female participants who are 21 to 80 years of age at the time of signing the informed consent.
* Participants with Canadian Cardiovascular Society (CCS) class III or IV chronic refractory angina.
* Participants without control of their angina symptoms in spite of maximal tolerated doses of anti-angina drugs. Participants must be on optimal therapy for their angina and must have been on a stable anti-anginal medication regimen for at least 4 weeks before signing the informed consent form.
* Participants with obstructive coronary disease unsuitable for conventional revascularization due to unsuitable anatomy or comorbidity as determined at the site and confirmed by an independent adjudication committee.
* Participants must have evidence of inducible myocardial ischemia.
* Participants must experience angina episodes.
* Participants must be able to complete 2 exercise tolerance tests on the treadmill within 3 weeks of randomization.
* If female of childbearing potential, subject must not be pregnant and agree to employ adequate birth control measures for the duration of the study.

Main Exclusion Criteria:

* Cardiovascular hospitalization within 60 days prior to potential study enrollment. Participant has had a successful or partially successful coronary artery bypass graft (CABG) within 6 months or PCTA within 60 days of potential study enrollment.
* Participant has had a placement of a bi-ventricular pacemaker for cardiac resynchronization therapy (CRT) for heart failure within 180 days of potential study enrollment.
* Participant has documented stroke or transient ischemic attacks (TIAs) within 60 days of potential study enrollment.
* Participant has a history of moderate to severe aortic stenosis; or severe aortic insufficiency; or severe mitral stenosis; or severe mitral insufficiency.
* Participant has a prosthetic aortic valve or a mechanical mitral valve replacement.
* Participant has severe co-morbidity associated with a reduction in life expectancy to less than 3 years as a result of chronic medical illnesses.
* Participants with cancer are excluded with the following exceptions:

  * Subjects with in-situ non-melanoma skin cancer or in-situ cervical cancer are not excluded.
  * Participants that have been cancer free for >= 5 years as determined by their oncologist are not excluded. Subjects with a prior history of stem cell transplant for cancer are excluded no matter how long they have been cancer-free.
* Participants with a history of leukemia or other bone marrow disease.
* Participant has sickle cell disease or sickle cell trait.
* Participants with proliferative retinopathy.
* Participants with Hb A1c > 9%.
* Participant has platelet counts >10% above the upper limit of normal (ULN) or platelet counts < 70,000.
* Participant has a hematocrit < 30% prior to potential study enrollment.
* Participant has a serum creatinine > 2.5 mg/dL prior to potential study enrollment.
* Participant tests positive for HIV, hepatitis B, or hepatitis C, or is on chronic immunosuppressive medications, or has had a previous stem cell transplant.
* Participant has a known contraindication to Neupogen (filgrastim) or G-CSF.
* Participant was previously enrolled in an active treatment group of cell therapy trials for cardiovascular disease including any phase of CD34+ stem cell trials.
* Left ventricular (LV) thickness of < 7 mm in the target areas of injection as measured by during a 2-D echocardiogram (ECHO).
* Atrial fibrillation, atrial flutter, or other uncontrolled arrhythmias that would prohibit accurate electromechanical mapping and NOGA-guided intramyocardial injection.
* Bleeding diathesis with an INR > 1.8 when not receiving anti-thrombotic therapy.
* Hepatic dysfunction as evidenced by elevated AST or ALT levels > 2.5 x ULN.
* Any previous transplant requiring immunosuppression.
* Disease state requiring chronic immunosuppression.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2012-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caladrius Study Director, Study Director — Caladrius Biosciences
Locations (41):
- United States (41):
  - Birmingham, Alabama
  - Gilbert, Arizona
  - Phoenix, Arizona
  - La Jolla, California
  - Los Angeles, California
  - Oxnard, California
  - San Diego, California
  - Stanford, California
  - Boynton Beach, Florida
  - Daytona Beach, Florida
  - Gainesville, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Chicago, Illinois
  - Iowa City, Iowa
  - Louisville, Kentucky
  - New Orleans, Louisiana
  - Boston, Massachusetts
  - Saginaw, Michigan
  - Minneapolis, Minnesota
  - Rochester, Minnesota
  - Haddon Heights, New Jersey
  - Newark, New Jersey
  - New York, New York
  - Charlotte, North Carolina
  - Durham, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Germantown, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Seattle, Washington
  - Madison, Wisconsin
  - Milwaukee, Wisconsin

REFERENCES:
- [Derived] Povsic TJ, Henry TD, Traverse JH, Fortuin FD, Schaer GL, Kereiakes DJ, Schatz RA, Zeiher AM, White CJ, Stewart DJ, Jolicoeur EM, Bass T, Henderson DA, Dignacco P, Gu Z, Al-Khalidi HR, Junge C, Nada A, Hunt AS, Losordo DW; RENEW Investigators. The RENEW Trial: Efficacy and Safety of Intramyocardial Autologous CD34(+) Cell Administration in Patients With Refractory Angina. JACC Cardiovasc Interv. 2016 Aug 8;9(15):1576-85. doi: 10.1016/j.jcin.2016.05.003. PMID 27491607
- [Derived] Povsic TJ, Junge C, Nada A, Schatz RA, Harrington RA, Davidson CJ, Fortuin FD, Kereiakes DJ, Mendelsohn FO, Sherman W, Schaer GL, White CJ, Stewart D, Story K, Losordo DW, Henry TD. A phase 3, randomized, double-blinded, active-controlled, unblinded standard of care study assessing the efficacy and safety of intramyocardial autologous CD34+ cell administration in patients with refractory angina: design of the RENEW study. Am Heart J. 2013 Jun;165(6):854-861.e2. doi: 10.1016/j.ahj.2013.03.003. Epub 2013 Apr 19. PMID 23708155

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started in May 2012 and completed in November 2015.
Pre-assignment Details: 291 participants provided informed consent and were screened. There were 179 screen failures. 112 participants were randomized and treated. Note that during treatment the number of arms increased from 3 to 4 to include "Not Injected" arm as 6 participants in Treatment and Active Control Arms did not have intramyocardial injections.
Groups:
- Active Control Arm: Targeted intramyocardial delivery of placebo after granulocyte-colony stimulating factor (G-CSF) mobilization and apheresis.
- Unblinded Standard of Care (SOC) Arm: No study-related procedures were performed.
- Not Injected Arm: Participants randomized into the Treatment Arm or Active Control Arm who did not undergo targeted intramyocardial delivery of 1 x 10^5 Auto-CD34+ cells or placebo, respectively.
Period: Randomization
Arm/Group | Treatment Arm | Active Control Arm | Unblinded Standard of Care (SOC) Arm | Not Injected Arm
Started | 57 | 27 | 28 | 0 (Participants not randomized into Not Injected arm, but some were re-assigned here during treatment.)
Completed | 57 | 27 | 28 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Treatment
Arm/Group | Treatment Arm | Active Control Arm | Unblinded Standard of Care (SOC) Arm | Not Injected Arm
Started | 50 | 28 | 28 | 6 (3 moved from Treatment (Tx) to Active Control (AC) Arm; 6 in Not injected Arm(4 from Tx ; 2 from AC))
Completed | 48 | 24 | 18 | 3
Not Completed | 2 | 4 | 10 | 3
Not completed — Death | 2 | 3 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 2 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 6 | 1
Not completed — Sponsor Decision | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Arms for baseline characteristics based on the Safety population as randomized i.e. randomized participants prior to treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm | Active Control Arm | Unblinded Standard of Care (SOC) Arm | Total
Number analyzed (Participants) | 57 | 27 | 28 | 112
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64 (8) | 64 (8) | 63 (10) | 64 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 4 | 18
  Male | 47 | 23 | 24 | 94

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total Exercise Time on Exercise Tolerance Test (ETT) Using the Modified Bruce Protocol
Description: Baseline (BL) is the average of the two total exercise times measured during the screening period.
Time Frame: Baseline and 12 month visit
Population: Participants in the Intent to Treat population defined as participants randomized to Treatment or Active Control arms. For participants not receiving intramyocardial injections, the missing values were imputed i.e. replaced with substituted values from the baseline.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Treatment Arm | Active Control Arm
Number analyzed (Participants) | 57 | 27
seconds | 108.7 (194.3) | 90.0 (184.7)

2. Secondary Outcome: Angina Frequency (Episodes Per Week) at the 12 Month Follow-up Visit
Description: Participants self-reported angina episodes utilizing an electronic diary for 4 weeks at baseline (screening period) and in the 4 weeks before the 3, 6 and 12 month follow-up visits.
Time Frame: Baseline and 12 month visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: angina episodes per week
Arm/Group | Treatment Arm | Active Control Arm
Number analyzed (Participants) | 57 | 27
angina episodes per week
  Number of weekly angina episodes at baseline | 20.1 (13.0) | 16.5 (9.4)
  Number of weekly angina episodes at Month 12 visit | 7.7 (9.5) | 5.4 (7.4)

3. Secondary Outcome: Change From Baseline in Total Exercise Time on Exercise Tolerance Test (ETT) at the 6 Month Follow-up Visit
Description: Baseline (BL) is the average of the two total exercise times measured during the screening period.
Time Frame: Baseline and 6 month visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Treatment Arm | Active Control Arm
Number analyzed (Participants) | 57 | 27
seconds | 126.5 (161.1) | 93.5 (138.6)

4. Secondary Outcome: Angina Frequency (Episodes Per Week) at the 6 Month Follow-up Visit
Time Frame: 6 month visit
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: angina episodes per week
Arm/Group | Treatment Arm | Active Control Arm
Number analyzed (Participants) | 57 | 27
angina episodes per week | 8.0 (9.6) | 8.4 (9.8)

5. Secondary Outcome: Percentage of Participants With Incidences of MACE From Randomization Until the End of the 24 Month Follow-up Period
Description: Major adverse cardiac events (MACE) defined as death, cardiac hospitalization, non-fatal myocardial infarction and stroke, as adjudicated by an independent clinical endpoint classification (CEC) committee.
  The category Total MACE includes death, cardiovascular hospitalization, myocardial infarction or stroke.
Time Frame: From randomization until the end of the 24 month follow-up period
Population: Participants in the safety population as Treated.
Measure: Number (95% Confidence Interval); unit: percent
Arm/Group | Treatment Arm | Active Control Arm | Unblinded Standard of Care (SOC) Arm | Not Injected Arm
Number analyzed (Participants) | 50 | 28 | 28 | 6
percent
  Cardiovascular Hospitalization | 42.0 [28.2 to 56.8] | 32.1 [15.9 to 52.4] | 64.3 [44.1 to 81.4] | 33.3 [4.3 to 77.7]
  Death | 4.0 [0.5 to 13.7] | 10.7 [2.3 to 28.2] | 7.1 [0.9 to 23.5] | 0 [0 to 0]
  Myocardial Infarction | 10.0 [3.3 to 21.8] | 10.7 [2.3 to 28.2] | 7.1 [0.9 to 23.5] | 33.3 [4.3 to 77.7]
  Stroke | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Total MACE (see outcome measure description) | 46.0 [31.8 to 60.7] | 42.9 [24.5 to 62.8] | 67.9 [47.6 to 84.1] | 33.3 [4.3 to 77.7]
  Myocardial Perforation | 4.0 [0.5 to 13.7] | 0 [0 to 0] | 0 [0 to 0] | 16.7 [0.4 to 64.1]
  Ventricular Arrhythmia | 2.0 [0.1 to 10.6] | 7.1 [0.9 to 23.5] | 3.6 [0.1 to 18.3] | 0 [0 to 0]

6. Secondary Outcome: Percentage of Participants With at Least One Serious Adverse Event (SAE) From Randomization Until the End of the 24 Month Follow-up Period
Time Frame: From randomization until the end of the 24 month follow-up period
Population: Safety Population as Treated.
Measure: Number; unit: percent
Arm/Group | Treatment Arm | Active Control Arm | Unblinded Standard of Care (SOC) Arm | Not Injected Arm
Number analyzed (Participants) | 50 | 28 | 28 | 6
percent | 62.0 | 60.7 | 78.6 | 50.0

ADVERSE EVENTS:
Time Frame: From randomization until the end of the 24 month follow-up period
Groups:
- Not Treated Arm: Participants randomized into the Treatment Arm or Active Control Arm who did not undergo targeted intramyocardial delivery of 1 x 10^5 Auto-CD34+ cells or placebo, respectively.
Arm/Group | Treatment Arm | Active Control Arm | Unblinded Standard of Care (SOC) Arm | Not Treated Arm
Serious Adverse Events (participants affected / at risk) | 31/50 | 17/28 | 22/28 | 3/6
Other Adverse Events (participants affected / at risk) | 48/50 | 26/28 | 23/28 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=50) | Active Control Arm (N=28) | Unblinded Standard of Care (SOC) Arm (N=28) | Not Treated Arm (N=6)
Angina pectoris (Cardiac disorders) | 7 (9) | 2 (3) | 11 (18) | 0 (0)
Angina unstable (Cardiac disorders) | 4 (7) | 2 (2) | 3 (3) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 3 (3) | 3 (3) | 1 (1) | 1 (2)
Cardiac failure congestive (Cardiac disorders) | 3 (4) | 2 (3) | 2 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronotropic incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery perforation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Sudden cardiac death (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device electrical impedance issue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocution (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular complication associated with device (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Intermittent claudication (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endocarditis bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Carotid sinus syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal infarction (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Brain neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningioma malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=50) | Active Control Arm (N=28) | Unblinded Standard of Care (SOC) Arm (N=28) | Not Treated Arm (N=6)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 3 (3) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 17 (26) | 11 (15) | 4 (4) | 2 (4)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 4 (5) | 2 (2) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (8) | 0 (0) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (4) | 2 (2) | 2 (3)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 7 (7) | 5 (6) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Chills (General disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 9 (9) | 8 (9) | 3 (3) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 5 (6) | 2 (4) | 6 (6) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Vessel puncture site haematoma (General disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 5 (6) | 4 (5) | 5 (7) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 3 (3) | 3 (3) | 0 (0)
Nasopharyngitis (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 9 (10) | 2 (2) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 13 (14) | 8 (13) | 2 (3) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (16) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Blood creatine phosphokinase MB increased (Investigations) | 4 (4) | 6 (6) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 5 (9) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Haematology test abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 4 (4) | 5 (5) | 0 (0) | 0 (0)
Prostatic specific antigen increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 3 (4) | 2 (2) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (12) | 11 (16) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (12) | 12 (14) | 5 (7) | 1 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 6 (8) | 2 (2) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 7 (7) | 2 (2) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 5 (6) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 6 (6) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 7 (7) | 5 (6) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 5 (6) | 1 (1)
Dizziness (Nervous system disorders) | 7 (8) | 7 (7) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 9 (10) | 5 (9) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 3 (3) | 2 (2) | 0 (0) | 2 (2)
Memory impairment (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Anxiety (Psychiatric disorders) | 3 (3) | 6 (6) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 3 (4) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (7) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 3 (3) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 5 (6) | 3 (3) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Study terminated early due to business considerations. Participants in Treatment or Active Control arms who did not have injection of target cells/placebo assigned to Not Injected Arm. Not included in efficacy analysis but in safety follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Baxalta's agreements with PIs may vary per requirements of individual PI, but contain common elements. For this study, results may not be published without prior written approval of Sponsor.